CLINICAL TRIAL: NCT04085510
Title: Improving Surveillance of Women With Personal History of Breast Cancer Using Contrast-Enhanced Mammography (CEM)
Brief Title: Tomosynthesis vs. Contrast-Enhanced Mammography in Women With Personal History of Breast Cancer in Western Pennsylvania
Acronym: TOCEM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wendie Berg (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Wendie Berg, Professor of Radiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY19060359
Record Dates: First submitted 2019-09-06; First posted 2019-09-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Female; Breast Cancer; Breast Neoplasms; Neoplasms
Keywords: breast cancer screening; digital breast tomosynthesis; contrast-enhanced mammogram
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Contrast-enhanced mammogram (Experimental): All women will receive both 3D mammography and contrast-enhanced mammography for breast cancer screening; the order of interpretation will vary for each of two radiologists
  Interventions: Device: Contrast-enhanced mammogram

INTERVENTIONS:
Device: Contrast-enhanced mammogram — Contrast-enhanced mammography (CEM) is a new FDA-approved exam that is similar to magnetic resonance imaging (MRI) in depicting breast cancers due to increased and leaky blood vessels. Contrast-enhanced mammography is used as an adjunct following mammography and/or ultrasound examinations to localize a known or suspected lesion.

SUMMARY:
This is a prospective clinical trial that will examine if contrast-enhanced mammography substantially improves breast cancer detection compared to mammography with tomosynthesis, with minimal increase in false-positives, in women with a personal history of breast cancer.

DETAILED DESCRIPTION:
The investigators expect to show in a prospective clinical trial that, in women with a personal history of breast cancer, contrast-enhanced mammography substantially improves breast cancer detection compared to mammography with tomosynthesis, with minimal increase in false positives. The investigators expect a substantial increase in node-negative invasive cancers in particular. Because DBT will be interpreted first by one reader, and CEM will be interpreted first, and independently, by a second reader, there will also be an assessment of performance of tomosynthesis alone or CEM alone in this population. Participants will be invited to three rounds of annual screening with CEM. CEM must be performed at the time of or within 6 weeks of routine annual mammogram with tomosynthesis.

ELIGIBILITY:
Inclusion Criteria:

-Asymptomatic women, ages 30-85, with a personal history of breast cancer who have had at least one routine mammogram since treatment.

Exclusion Criteria:

* Women with a history of prior iodinated contrast reaction
* Women with implant(s) in the breasts to be screened (as this creates artifacts and diagnostic performance of imaging in women with implants likely does not generalize to those without implants, and the sample size with implants would be too small to infer conclusions)
* Women who have had bilateral mastectomy
* Women with a history of kidney failure or estimated glomerular filtration rate (eGFR) < 30 mL/min
* Pregnancy or lactation
* Women actively being treated for cancer of any type with chemotherapy
* Lump or other breast symptoms
* Abnormality on prior breast imaging that is being followed.

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1647 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Cancer Detection | 48 months
  Number of participants with cancer detected with contrast-enhanced mammography compared to tomosynthesis. Number of patients recalled for additional testing by each imaging test who do not have cancer (false positives). Outcomes will be assessed for both prevalence and incidence screens.

SECONDARY OUTCOMES:
Reader Validation | 48 months
  Reader validation will be performed at study conclusion: number of cancers detected with contrast-enhanced mammography or tomosynthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Wendie Berg, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Magee Womancare Passavant Cranberry, Cranberry Township, Pennsylvania
  - Magee Womancare Monroeville, Monroeville, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Images may be shared with secondary investigators, including commercial companies after removal of all identifiers. All participant identification (name, patient number, birth date) will be removed prior to sharing.
Supporting Information: Study Protocol
Time Frame: At study conclusion
Access Criteria: Participant imaging may be shared with secondary investigators, including commercial companies either by electronic transfers or via disc downloads. All participant identification will be removed prior to the images release.